CLINICAL TRIAL: NCT04902248
Title: Endoscopic Application of Over-the-scope Clips (OTSC) vs. Angiographic Embolization in Patients With Refractory Non-variceal Upper Gastrointestinal Bleeding: a Multicenter Randomized Comparison
Brief Title: OTSC vs. Angiographic Embolization in Patients With Refractory Non-variceal Upper Gastrointestinal Bleeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OTSCTAE
Record Dates: First submitted 2021-05-14; First posted 2021-05-26 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: Over-the-scope clips; angiographic embolization
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Over-the-scope clips (Experimental): The OTSC® System Set is an instrument for flexible endoscopy
  The OTSC® System Set consists of an applicator cap with a mounted OTSC® clip, thread, thread retriever and a hand wheel for clip release.
  The OTSC® clip is delivered by means of an applicator cap mounted to the tip of gastroscopes or colonoscopes. The clip is released by tightening the thread with the hand wheel.
  The OTSC® clip for flexible endoscopy is a superelastic Nitinol device for compression and approximation of tissue in the digestive tract
  Interventions: Device: The OTSC® System Set
- angiographic embolization (Experimental): The procedure was performed in the angiographic suite and under local anaesthetics to the patient's groin. The celiac and then gastroduodenal artery or the left gastric artery was selectively cannulated depending on ulcer location.
  Coils were deposited distal to the bleeding point. Gel foam particles were then packed into the artery and its collaterals. This was followed by further coils deposited in its proximal portion until complete cessation of arterial flow. Our protocol requested empiric embolisation of the artery even in the absence of active contrast extravasation or a pseudoaneurysm.
  Interventions: Procedure: angiographic embolization

INTERVENTIONS:
Device: The OTSC® System Set — The endoscope was extracted and equipped with the OTSC system. OTSC system is deployed on the lesion with suction to target lesion
  Arms: Over-the-scope clips
Procedure: angiographic embolization — Transcatheter selective embolization to bleeding arteries
  Arms: angiographic embolization

SUMMARY:
In the management of patients with acute upper non-variceal upper gastrointestinal bleeding, further bleeding is the most important adverse factor predictive of mortality. In the United Kingdom Audit on acute upper gastrointestinal bleeding, clinical evidence of further bleeding was reported in 13% of patients following the first endoscopy and 27% of them died. The use of OTSC has emerged as an alternative before angiographic embolization(TAE) which is often considered most definitive.

We propose to define the algorithm in the management of patients with refractory bleeding from their peptic ulcers or other non variceal causes. We hypothesize that endoscopic use of OTSC compares favourably with TAE and both lead to similar outcomes. An equivalence of the two modalities may mean that endoscopic application of OTSC should be attempted before TAE as often we need to document further bleeds with endoscopy and a second treatment should be instituted at the same time.

DETAILED DESCRIPTION:
The current standard of care in patients with refractory bleeding from their peptic ulcers and other non-variceal causes has not been defined. An International Consensus Group recommends a surgical consult when endoscopic treatment has failed and TAE should be considered as an alternative. The European guidelines recommend the use of either surgery or angiographic embolization. There has not been a fully published RCT that compares angiographic treatment to surgery in those with refractory bleeding. Several comparative series mostly retrospective and their meta-analyses suggest that outcomes following TAE would not be dissimilar to those after surgery. Common to these reports, TAE is associated with a higher rate of further bleeds. In our meta-analysis , the pooled rate of further bleeds after TAE was 51/178(32%) compared to that of 26/241 (14.9%) after surgery. A high rate of further bleeding can be understood because of a rich vascular supply to peptic ulcers especially those in the bulbar duodenum. A bulbar ulcer receives dual arterial supply from celiac and superior mesenteric arteries. Embolization to these arteries can therefore be challenging. In a population-based study from northern Europe that included 282 patients (97 TAE and 185 surgery), the overall hazard of deaths after TAE decreased by 1/3 when compared to surgery. Many argue that TAE is preferred over surgery in the algorithm of management.

The use of OTSC has emerged as an alternative before TAE which is often considered most definitive. A multicenter randomized controlled trial that compared OTSC and standard endoscopic treatment mostly through-the-scope clips in patients with refractory bleeding peptic ulcers; 66 patients were randomized and control of bleeding over 30 days was better with the use of OTSC (15.2% vs. 57.6%). A Mayo Clinic group reported OTSC treatment in 67 high risk lesions defined by those near an arterial complex (bulbar or angular/lesser curve ulceration) with an artery larger than 2 mm, deep excavated fibrotic ulcer with major stigmata and those that failed standard endoscopic therapy (through-the-scope clips and/or thermal device); 47 (70.1%) remained free of further bleeds at day 30 10.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients presented with overt signs of acute upper gastrointestinal bleeding (hematemesis, melena and/or hypotension) 2. documented bleeding lesion at endoscopy (ulcer, dieulafoy's lesion and others), further bleeds (persistent or recurrent) after endoscopic hemostasis (thermal or hemoclips) as defined by an International Consensus Group

Exclusion Criteria:

1. without a full informed consent from the patient or his next of kin
2. Age <18 years
3. Pregnant
4. Lactating women
5. patients with known allergy to intravenous contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2021-11-27 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
further bleeding | within 30 days after randomization
  Further bleeding is a composite of persistent or recurrent bleeding. Persistent bleeding is defined by active bleeding that cannot be stopped despite study intervention. For assessment of treatment efficacy, a repeat endoscopy can be performed to document further bleeding (fresh blood in the stomach and active bleeding or major stigmata of bleeding to the previously treated lesion).

SECONDARY OUTCOMES:
further interventions | within 30 days after randomization
  repeat endoscopic therapy, interventional radiology or surgery performed for management of further bleeds or a complication of a study intervention
blood transfusion | within 30 days after randomization
  total units of blood transfusion
length of hospitalization | within 30 days after randomization
  duration of hospitalization
length of ICU stay | within 30 days after randomization
  duration of ICU stay
mortality related to bleeding | within 30 days after randomization
  the number of bleeding caused death
all cause mortality | within 30 days after randomization
  the number of death

CONTACTS AND LOCATIONS:
Overall Officials: Yau Wong James Lau, MD, Principal Investigator — The Chinese University of HongKong
Locations (5):
- China (3):
  - Beijing friendship Hospital, Beijing, Beijing Municipality
  - the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Huaxi Hospital of Sichuan University, Chengdu, Sichuan
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, N.T., Hong Kong
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barkun AN, Almadi M, Kuipers EJ, Laine L, Sung J, Tse F, Leontiadis GI, Abraham NS, Calvet X, Chan FKL, Douketis J, Enns R, Gralnek IM, Jairath V, Jensen D, Lau J, Lip GYH, Loffroy R, Maluf-Filho F, Meltzer AC, Reddy N, Saltzman JR, Marshall JK, Bardou M. Management of Nonvariceal Upper Gastrointestinal Bleeding: Guideline Recommendations From the International Consensus Group. Ann Intern Med. 2019 Dec 3;171(11):805-822. doi: 10.7326/M19-1795. Epub 2019 Oct 22. PMID 31634917
- [Result] Gralnek IM, Dumonceau JM, Kuipers EJ, Lanas A, Sanders DS, Kurien M, Rotondano G, Hucl T, Dinis-Ribeiro M, Marmo R, Racz I, Arezzo A, Hoffmann RT, Lesur G, de Franchis R, Aabakken L, Veitch A, Radaelli F, Salgueiro P, Cardoso R, Maia L, Zullo A, Cipolletta L, Hassan C. Diagnosis and management of nonvariceal upper gastrointestinal hemorrhage: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2015 Oct;47(10):a1-46. doi: 10.1055/s-0034-1393172. Epub 2015 Sep 29. PMID 26417980
- [Result] Kyaw M, Tse Y, Ang D, Ang TL, Lau J. Embolization versus surgery for peptic ulcer bleeding after failed endoscopic hemostasis: a meta-analysis. Endosc Int Open. 2014 Mar;2(1):E6-E14. doi: 10.1055/s-0034-1365235. Epub 2014 Mar 7. PMID 26134614
- [Result] Beggs AD, Dilworth MP, Powell SL, Atherton H, Griffiths EA. A systematic review of transarterial embolization versus emergency surgery in treatment of major nonvariceal upper gastrointestinal bleeding. Clin Exp Gastroenterol. 2014 Apr 16;7:93-104. doi: 10.2147/CEG.S56725. eCollection 2014. PMID 24790465
- [Result] Tarasconi A, Baiocchi GL, Pattonieri V, Perrone G, Abongwa HK, Molfino S, Portolani N, Sartelli M, Di Saverio S, Heyer A, Ansaloni L, Coccolini F, Catena F. Transcatheter arterial embolization versus surgery for refractory non-variceal upper gastrointestinal bleeding: a meta-analysis. World J Emerg Surg. 2019 Feb 1;14:3. doi: 10.1186/s13017-019-0223-8. eCollection 2019. PMID 30733822
- [Result] Sverden E, Mattsson F, Lindstrom D, Sonden A, Lu Y, Lagergren J. Transcatheter Arterial Embolization Compared With Surgery for Uncontrolled Peptic Ulcer Bleeding: A Population-based Cohort Study. Ann Surg. 2019 Feb;269(2):304-309. doi: 10.1097/SLA.0000000000002565. PMID 29064894
- [Result] Schmidt A, Golder S, Goetz M, Meining A, Lau J, von Delius S, Escher M, Hoffmann A, Wiest R, Messmann H, Kratt T, Walter B, Bettinger D, Caca K. Over-the-Scope Clips Are More Effective Than Standard Endoscopic Therapy for Patients With Recurrent Bleeding of Peptic Ulcers. Gastroenterology. 2018 Sep;155(3):674-686.e6. doi: 10.1053/j.gastro.2018.05.037. Epub 2018 May 24. PMID 29803838